CLINICAL TRIAL: NCT06511206
Title: Determination of the Optimal Nutrient Mix to Acutely Increase Plasma Ketones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NL86023.068.23
Record Dates: First submitted 2024-06-20; First posted 2024-07-19 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-10

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — 5,11-methenyltetrahydrohomofolate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 25g MCT-based nutrient mix (Experimental)
  Interventions: Dietary Supplement: 25g MCT-based nutrient mix
- 25g MCT-based nutrient mix + cofactors (Experimental)
  Interventions: Dietary Supplement: 25g MCT-based nutrient mix + cofactors
- non-ketogenic control (Placebo Comparator)
  Interventions: Dietary Supplement: non-ketogenic control

INTERVENTIONS:
Dietary Supplement: 25g MCT-based nutrient mix — The 25g MCT-based nutrient mix will be consumed two hours after breakfast.
  Arms: 25g MCT-based nutrient mix
Dietary Supplement: 25g MCT-based nutrient mix + cofactors — The 25g MCT-based nutrient mix + cofactors will be consumed two hours after breakfast.
  Arms: 25g MCT-based nutrient mix + cofactors
Dietary Supplement: non-ketogenic control — The non-ketogenic control will be consumed two hours after breakfast.
  Arms: non-ketogenic control

SUMMARY:
This study will be performed to determine the optimal nutrient mix (predominantly based on medium-chain triglycerides (MCTs)) to induce a mild ketogenic state in healthy older (60-80y), overweight/obese (BMI: 25-35 kg/m2) individuals. Since the aim is to induce a mild ketogenic state, a 25g MCT-based nutrient mix, a 25g MCT-based nutrient mix + cofactors, or a non-ketogenic control will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60-80 years
* Body mass index (BMI) 25-35 kg/m2
* Stable dietary habits (no weight loss or gain > 5 kg in the past 3 months)
* Participants are able to provide signed and dated written informed consent prior to any study specific procedures

Exclusion Criteria:

* Type 2 diabetes
* Pre-diabetes based on one or a combination of the following criteria:

  * ImpairedFastingGlucose(IFG):Fasting plasma glucose ≥ 6.1mmol/l and ≤ 6.9 mmol/l.
  * HbA1c of 5.7-6.4%.
* Participants with active congestive heart failure and/or severe renal and or liver insufficiency
* Uncontrolled hypertension
* Alcohol consumption of > 3 servings per day for man and > 2 servings per day for woman
* Unstable body weight (weight gain or loss > 5 kg in the last 3 months)
* Previous enrolment in a clinical study with an investigational product during the last 3 months or as judged by the investigator which would possibly hamper our study results
* Significant food allergies/intolerance (seriously hampering study meals)
* Participants who do not want to be informed about unexpected medical findings
* Blood donation during or within 2 months prior to the study

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Plasma ketone levels | Testday 1, 2, and 3
  The primary outcome is plasma ketone levels determined regularly over a defined time period after ingestion of the respective nutritional supplements, expressed as area under the curve (AUC).

OTHER OUTCOMES:
Whole-body fat oxidation | Testday 1, 2, and 3
  An exploratory outcome is the whole-body fat oxidation / substrate utilization determined regularly over a defined time period after ingestion of the respective nutritional supplements, expressed as g/min and respiratory exchange ratio.
Energy expenditure | Testday 1, 2, and 3
  An exploratory outcome is the energy expenditure determined regularly over a defined time period after ingestion of the respective nutritional supplements, expressed as kJ/min.
Metabolites in the blood | Testday 1, 2, and 3
  An exploratory outcome is the plasma metabolite levels determined regularly over a defined time period after ingestion of the respective nutritional supplements, expressed as i.e. glucose in mmol/L, insulin in pmol/L.
Interstitial ketone levels | Testday 1, 2, and 3
  An exploratory outcome is the interstitial ketone levels determined regularly over a defined time period after ingestion of the respective nutritional supplements, expressed as μM.

CONTACTS AND LOCATIONS:
Overall Officials: Joris Hoeks, Dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No